CLINICAL TRIAL: NCT02347982
Title: Epidemiology of Cardiovascular Disease in Elderly Turkish Population
Acronym: ELDER-TURK
Status: Completed | Type: Observational
Sponsor: Turkish Society of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: ELDER-TURK
Record Dates: First submitted 2015-01-20; First posted 2015-01-28 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Diseases
Keywords: Turkey; Epidemiologic
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will compose a national database of cardiovascular diseases' risk factors, concomitant diseases and the drug usage among the elderly patients in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* patients signed patient informed sheet and informed consent form
* patients ≥65 years old
* patients followed-up cardiology clinics

Exclusion Criteria:

* patients under 65 years old

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥65 years followed-up at cardiology clinics
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To generate a national database for cardiovascular diseases for elderly patients in Turkey | [Recruited and could be analysed at least 2500 patients after 9 months]

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Zoghi, Prof, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Medicine, Izmir, Turkey (Türkiye)